CLINICAL TRIAL: NCT03049189
Title: A Prospective, Randomised, Controlled, Open-label, Multicentre Phase III Study to Evaluate Efficacy and Safety of Peptide Receptor Radionuclide Therapy (PRRT) With 177Lu-Edotreotide Compared to Targeted Molecular Therapy With Everolimus in Patients With Inoperable, Progressive, Somatostatin Receptor-positive (SSTR+), Neuroendocrine Tumours of Gastroenteric or Pancreatic Origin (GEP-NET)
Brief Title: Efficacy and Safety of 177Lu-edotreotide PRRT in GEP-NET Patients
Acronym: COMPETE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ITM Solucin GmbH (Industry)
Collaborators: ABX CRO (Other); PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITM-LET-01
Record Dates: First submitted 2017-01-13; First posted 2017-02-09 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors
Keywords: non-functional and functional P-NET; non-functional GE-NET
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-; Everolimus; amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 177Lu-edotreotide PRRT (Experimental): 177Lu-edotreotide (177Lu-DOTATOC)
  A maximum of four cycles of 7.5 ± 0.7 GBq (gigabequerel) 177Lu-edotreotide, each.
  Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 4 cycles, 90 days apart (total duration: 270 days/9 months)
  Interventions: Drug: 177Lu-edotreotide PRRT; Other: Amino-Acid Solution
- Everolimus (Active Comparator): Everolimus (Afinitor ®)
  Doses: 10 mg/d Route of administration: Oral Duration of treatment: Continuous daily treatment until diagnosis of progression or End of Study (EOS)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: 177Lu-edotreotide PRRT — PRRT using 177Lu-edotreotide will be performed 3-monthly. A maximum of four cycles will be administered.
  Other Names: 177Lu-DOTATOC; 177Lu-Edo
  Arms: 177Lu-edotreotide PRRT
Drug: Everolimus — Everolimus will be administered as a standard dosis of 10 mg daily which may be reduced where required for acceptable tolerability.
  Other Names: Afinitor
  Arms: Everolimus
Other: Amino-Acid Solution — The Amino-Acid Solution (AAS) to be used in this study will contain a mixture of 25 g lysine and 25 g arginine diluted in 2000 mL of electrolyte solution, infused over 4 - 6 h, starting 30 - 60 min before PRRT
  Other Names: Arginine-Lysine Solution
  Arms: 177Lu-edotreotide PRRT

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of Peptide Receptor Radionuclide Therapy (PRRT) with 177Lu-Edotreotide compared to targeted molecular therapy with Everolimus in patients with inoperable, progressive, somatostatin receptor-positive (SSTR+), neuroendocrine tumours of gastroenteric or pancreatic origin (GEP-NET).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of well-differentiated neuro-endocrine tumour of non-functional gastroenteric origin (GE-NET) or both functional or non-functional pancreatic origin (P-NET)
* Measurable disease per RECIST 1.1
* Somatostatin receptor positive (SSTR+) disease
* Progressive disease based on RECIST 1.1. criteria as evidenced by two morphological imaging examinations made with the same imaging method (either CT or MRI)

Exclusion Criteria:

* Known hypersensitivity to edotreotide or everolimus
* Known hypersensitivity to DOTA, lutetium-177, or any excipient of edotreotide or everolimus or any other Rapamycin derivative
* Prior exposure to any peptide receptor radionuclide therapy (PRRT)
* Prior therapy with mTor inhibitors
* Prior EFR (external field radiation) to GEP-NET lesions within 90 days before randomisation or radioembolisation therapy
* Therapy with an investigational compound and/or medical device within 30 days prior to randomisation
* Indication for surgical lesion removal with curative potential
* Planned alternative therapy (for the period of study participation)
* Serious non-malignant disease
* Clinically relevant renal, hepatic, cardiovascular, or haematological organ dysfunction, potentially interfering with the safety of the study treatments
* Pregnant or breast-feeding women
* Subjects not able to declare meaningful informed consent on their own (e.g. with legal guardian for mental disorders) or any other vulnerable population to that sense (e.g. persons institutionalised, incarcerated etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 12 weeks +/- 14 days, up to 30 months
  PFS will be assessed individually per patient from date of randomization until the date of first documented progression or death, assessed up to 30 months, primary outcome will be measured by CT/MRI every 12 weeks +/- 14 days

SECONDARY OUTCOMES:
objective response rates (ORR) | 12 weeks +/- 14 days, up to 30 months
  ORR will be assessed, defined as the proportion of patients achieving partial response (PR) or complete response (CR) as best outcome, after treatment with 177Lu-edotreotide compared to everolimus
overall survival (OS) | 12 weeks +/- 14 days, up to 90 months
  OS as secondary outcome measure will be assessed per patient from date of randomization until the date of death

CONTACTS AND LOCATIONS:
Locations (52):
- United States (6):
  - Banner Health d.b.a. Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Stanford University, Stanford, California
  - Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Excel Diagnostics & Nuclear Oncology Center, Houston, Texas
- Australia (4):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Olivia Newton-John Cancer & Wellness Centre, Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Allgemeines Krankenhaus Wien, Vienna, Austria
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Czechia (2):
  - University Hospital Olomouc, Olomouc
  - University Hospital Motol, Prague
- France (6):
  - Hospices civils de Lyon, Bron
  - Centre Jean Perrin, Clermont-Ferrand
  - HP Hôpital Beaujon, Clichy
  - Institut de Recherche en Cancérologie de Montpellier (IRCM), Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - IUCT-Oncopole, Toulouse
- Germany (11):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - University Medical Center, Abteilung für Nuklearmedizin, Hamburg
  - Universitätsklinikum Magdeburg A.ö.R., Otto-von-Guericke Universität, Magdeburg
  - Philipps Universität Marburg, Marburg
  - Klinikum rechts der Isar Technische Universität München, Munich
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Italy (3):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) Srl, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - European Institute of Oncology (EIO), Milan
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands
- Poland (2):
  - MSC Memorial Cancer Centre, Gliwice
  - "Gammed" Izabela Chuchrowksa, Warsaw
- South Africa (2):
  - University Cape Town (UCT), Groote Schuur Hospital, Cape Town
  - University of Pretoria & Steve Biko Academic Hospital, Pretoria
- Spain (6):
  - Vall d'Hebron University Hospital, Barcelona
  - ICO Hospitalet, Granvia de l'Hospitalet, Barcelona
  - MD Anderson Cancer Center Madrid, Madrid
  - University Hospital 12 de Octubre, Madrid
  - Central University Hospital de Asturias (HUCA), Oviedo
  - University and Polytechnic Hospital La Fe, Valencia
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Inselspital, Universitätsspital Bern, Bern
  - UniversitätsSpital Zürich, Zurich
- United Kingdom (3):
  - Royal Free NHS Foundation Trust, London
  - Kings College Hospital, London
  - The Christie NHS Foundation Trust, Manchester